CLINICAL TRIAL: NCT02903394
Title: Coherence Imaging of the Cervical Epithelium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Jacobi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00070555; R01CA167421 (NIH)
Record Dates: First submitted 2016-09-01; First posted 2016-09-16 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Cervical Epithelia

ARMS (1):
- mLCI imaging (Experimental): mLCI device images cervical epithelium
  Interventions: Device: mLCI Device

INTERVENTIONS:
Device: mLCI Device — imaging of cervical epithelium using mLCI device

SUMMARY:
The purpose of this study is to develop a multiplexed low coherence interferometry (mLCI) endoscopic probe for mapping the epithelial types of the cervix. This vaginal mLCI probe will obtain optical measurements from the cervix. These measurements can be used to create a map of the surface cells that distinguishes ectocervical epithelia, endocervical epithelia, and the squamocolumnar junction (t-zone), which is the region where cervical dysplasia is most likely to occur.

ELIGIBILITY:
Inclusion Criteria:

* able to provide informed consent
* willing to abstain from sexual intercourse for at least 24 hours before study visit

Exclusion Criteria:

* pregnant
* using an intrauterine device (IUD)
* have a current gynecological infection or discharge
* have had any cervical surgery
* had medical or cosmetic surgery involving the reproductive organs or genitals within the past 6 months
* currently enrolled in any research studies involving the application of vaginal formulations
* employed or supervised by the study investigators
* have any other condition, that, in the opinion of the study clinician, would contraindicate participation in the study

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2017-10-24 (Actual); Study Completion 2017-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Wax, Ph.D., Principal Investigator — professor
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- mLCI Imaging (Pilot): Pilot study. 5 women from ages 24 to 34 recruited at Duke University (Durham, NC). Exclusion criteria included history of cervical dysplasia or previous surgery on the cervix, complaint of vaginal discharge or suspicion of sexually transmitted infection at the time of presentation, or positive urine pregnancy test.
- mLCI Imaging (Jacobi): Primary arm of present study. 50 women from ages 18 to 42 recruited from routine care population at New York City Health + Hospitals / Jacobi (Bronx, New York, NY). Exclusion criteria included history of cervical dysplasia or previous surgery on the cervix, complaint of vaginal discharge or suspicion of sexually transmitted infection at the time of presentation, or positive urine pregnancy test.
  Women were examined by speculum to visualize the cervix. Wallach colposcope was used to acquire a photograph of the cervix. mLCI probe was then inserted through speculum and placed against the cervix by endoscopic visual guidance provided through the probe. Optical interferometric data was acquired within a 20 mm field of view, and results were analyzed to determine tissue type.
Period: Overall Study
Arm/Group | mLCI Imaging (Pilot) | mLCI Imaging (Jacobi)
Started | 5 | 50
Completed | 5 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | mLCI Imaging (Pilot) | mLCI Imaging (Jacobi) | Total
Number analyzed (Participants) | 5 | 50 | 55
Age, Continuous [Mean (Full Range); unit: years] | 29.8 [24 to 34] | 29.4 [18 to 42] | 29.4 [18 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 50 | 55
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 16 | 16
  Not Hispanic or Latino | 5 | 34 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 26 | 28
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 16 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Interferometric Data Acquired From Cervical Epithelium
Description: measured by: ability to receive interferometric data from at least one portion of the cervical epithelium
Time Frame: day 1
Measure: Number; unit: patients
Arm/Group | mLCI Imaging (Pilot) | mLCI Imaging (Jacobi)
Number analyzed (Participants) | 5 | 50
patients | 3 | 41

2. Secondary Outcome: Number of Patients With Automated Classification of Cervical Epithelium
Description: The number of patients for which an interferometric tissue classification was made using optical mLCI data
Time Frame: day 1
Population: Patients from whom epithelial interferometric data were successfully captured and for whom a corresponding colposcope image could be registered. No pilot study patients were included as no colposcopic examination was conducted in the pilot phase.
Measure: Number; unit: patients
Groups:
- mLCI Imaging (Pilot): Pilot study. 5 women from ages 24 to 34recruited at Duke University (Durham, NC). Exclusion criteria included history of cervical dysplasia or previous surgery on the cervix, complaint of vaginal discharge or suspicion of sexually transmitted infection at the time of presentation, or positive urine pregnancy test.
Arm/Group | mLCI Imaging (Pilot) | mLCI Imaging (Jacobi)
Number analyzed (Participants) | 0 | 41
patients |  | 36

3. Secondary Outcome: Number and Frequency of Adverse Events
Description: Number of adverse events experienced by patients during the mLCI study.
Time Frame: day 1
Measure: Number; unit: events
Arm/Group | mLCI Imaging (Pilot) | mLCI Imaging (Jacobi)
Number analyzed (Participants) | 5 | 50
events | 0 | 0

ADVERSE EVENTS:
Time Frame: Day of study only
Arm/Group | mLCI Imaging (Pilot) | mLCI Imaging (Jacobi)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/50
Other Adverse Events (participants affected / at risk) | 0/5 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-17): https://cdn.clinicaltrials.gov/large-docs/94/NCT02903394/Prot_SAP_000.pdf